CLINICAL TRIAL: NCT05121012
Title: Molecular Imaging of Synaptic Loss in Multiple System Atrophy (MSA)
Brief Title: Synaptic Loss in Multiple System Atrophy
Status: Recruiting | Type: Observational
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Other Study IDs: 1920/15
Record Dates: First submitted 2021-09-29; First posted 2021-11-16 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Multiple System Atrophy; Progressive Supranuclear Palsy (PSP)
Keywords: Neurodegeneration; Positron Emission Tomography; Multiple System Atrophy; Biomarkers; Progressive Supranuclear Palsy
MeSH Terms: conditions — Multiple System Atrophy; Supranuclear Palsy, Progressive; Nerve Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood will be collected for analysis of inflammatory biomarkers (including CRP, IL-6, IL-1b, TNF, ferritin, ESR, NfL) and for storage in biobanks for future ethically approved studies.
  Cerebrospinal fluid (CSF) will be collected for analysis of cell count and for biomarkers (for MSA only).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with MSA: Patients with a diagnosis of MSA and either a clinical form MSA-C or MSA-P
  Interventions: Other: Study procedures for MSA patients
- Patients with Progressive Supranuclear Palsy: Patients with a diagnosis of PSP, either the clinical forms PSP-RS or PSP-P
  Interventions: Other: Study procedures for PSP patients

INTERVENTIONS:
Other: Study procedures for MSA patients — The group of MSA patients will undergo a collection of demographic data, a neurological examination with administration of clinical scales relevant for MSA, and a collection of venous blood sample for routine and biomarker analyses.
  Participants will undergo one PET scan with the tracer [11C]UCB-J, and one PET scan with the tracer [18F]FDG. All participants will also undergo one MRI scan.
  Participants will also undergo one lumbar puncture (optional).
  All procedures will be performed at baseline and after one-year follow-up.
  A subgroup of patients with MSA will also undergo, at one time point only, one PET scan with the tracer [18F]APN107.
  Groups: Patients with MSA
Other: Study procedures for PSP patients — The group of PSP patients will undergo a collection of demographic data, a neurological examination with administration of clinical scales relevant for PSP, and a collection of venous blood sample for routine and biomarker analyses. Participants will undergo one PET scan with the tracer [18F]APN107 and one MRI scan. All procedures will be performed at baseline and after one-year follow-up.
  Groups: Patients with Progressive Supranuclear Palsy

SUMMARY:
In this study the investigators would like to investigate the degree of damage of the synapses, an important part of the neurons vital for the communications between neurons, in Multiple System Atrophy (MSA), and pathology related to abnormal accumulation of a protein named tau, in Progressive Supranuclear Palsy (PSP).

DETAILED DESCRIPTION:
Multiple System Atrophy (MSA) is a chronic and progressive neurological disease, for which unfortunately there is no cure yet. It is known from pathological studies that the synapses (the terminal parts of the neurons) are affected in this disease, but the investigators don't know how, and how much this happens. An imaging tool called Positron Emission Tomography (PET) can study the integrity of the synapses by the use of a dedicated tracer, called [11C]UCB-J. In this study the investigators would like to study how, and how early, the synapse deteriorate in patients with MSA.

For this study, patients with the MSA will be enrolled. Participants will be asked to undergo a clinical visit with questionnaires and scales for motor and cognitive symptoms. Then, participants will come for a [11C]UCB-J PET scan, a [18F]FDG PET scan, to check the metabolism of the brain, and a MRI scan, to help the analysis of the PET. The participants will also be asked to perform a Lumbar puncture for a cerebrospinal fluid draw. This procedure will be optional.

A subgroup of up to 10 patients with MSA who took part to the main study will also undergo an imaging substudy, with a PET scan (only at a single timepoint) with the tracer [18F]APN107. [18F]APN107 is a novel tracer measuring a protein in the brain named tau. Tau abnormally accumulates in patients with a disease named Progressive Supranuclear Palsy (PSP) but not in MSA. It is sometimes very challenging to distinguish MSA and PSP on the basis of the clinical observation. We hope that a PET scan with [18F]APN107 could help distinguish these disorders more. This subgroup of patients with MSA will be compared with a group of up to 16 patients with PSP (the clinical forms named PSP-RS and PSP-P) who will undergo the following activities:

At baseline, a clinical visit with administration of pen-and-paper tests and scales,, a venous blood collection, an MRI scan and one [18F]APN107 PET scan; After approximately one year from baseline (follow-up), the repetition of the same activities as at baseline.

The results will help in understanding better the mechanisms underlying thiese two conditions and open new avenues for its treatment.

ELIGIBILITY:
Inclusion Criteria

MSA group:

Male or female, aged 45-80 at the time of informed consent. Meet criteria for diagnosis of probable or possible MSA (Gilman et al., 2008) (Appendix 1).

A female subject is eligible to participate if she is a) of non-childbearing potential, defined as pre-menopausal females with a documented tubal ligation or hysterectomy, or postmenopausal defined as 12 months of spontaneous amenorrhea or b) of childbearing potential but not pregnant (as determined by urinary pregnancy test on screening and on each study day), is not lactating and is willing to use one of the contraception methods listed below:

* Combined (estrogen and progesterone containing) hormonal contraception associated with initiation of ovulation( oral, intravaginal, or transdermal);
* Progesterone-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable);
* Intrauterine device;
* Intrauterine hormone releasing system;
* Bilateral tubal occlusion;
* Vasectomized partner;
* Sexual abstinence.

Male subject with a female partner of child-bearing potential must use one of the following contraceptive methods for 90 days after each dose of radiotracer:

* Condom plus partner use of a highly effective contraceptive (see point above) OR
* Abstinence Subjects must understand the nature of the study and be able to provide signed and dated written informed consent in accordance with local regulations before the conduct of any study-related procedures. They must be able and willing to participate in all scheduled evaluations, abide by all study restrictions, and complete all required tests and procedures.

Must have anticipated survival of ≥3 years (in the opinion of the Investigator).

Medical treatment of MSA and co-morbid medical conditions must be stable for at least 30 days prior to screening and between screening and baseline PET scan. Intermittently administered treatment may be considered stable if the dose and dosing frequency have been unchanged for the greater of 30 days or three dosing inbiomartervals (e.g. a treatment given once a month must be at a stable dose and dosing frequency for 3 months).

For inclusion in optional CSF sampling, written informed consent must be provided, either by separate signed and dated written informed consent or by specific written acknowledgement on the main study informed consent form, according to local procedure. Failure to participate in optional CSF sampling will have no influence on the subject's ability to participate in the main study.

In the opinion of the investigator, the subject must be considered likely to comply with the study protocol and to have high probability of completing the study.

PSP Group:

Male or female, aged 45-80 at the time of informed consent. Meet criteria for diagnosis of suggestive, probable or possible PSP - with preference for PSP-RS, PSP-OM, PSP-PI, PSP with gait freezing, and PSP-SL and PSP-P subtypes (Höglinger et al., 2017 (Appendix 2).

A female subject is eligible to participate if she is a) of non-childbearing potential, defined as pre-menopausal females with a documented tubal ligation or hysterectomy, or postmenopausal defined as 12 months of spontaneous amenorrhea or b) of childbearing potential but not pregnant (as determined by urinary pregnancy test on screening and on each study day), is not lactating and is willing to use one of the contraception methods listed below:

* Combined (estrogen and progesterone containing) hormonal contraception associated with initiation of ovulation( oral, intravaginal, or transdermal);
* Progesterone-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable);
* Intrauterine device;
* Intrauterine hormone releasing system;
* Bilateral tubal occlusion;
* Vasectomized partner; Sexual abstinence.

Male subject with a female partner of child-bearing potential must use one of the following contraceptive methods for 90 days after each dose of radiotracer:

• Condom plus partner use of a highly effective contraceptive (see point above) OR Abstinence Subjects must understand the nature of the study and be able to provide signed and dated written informed consent in accordance with local regulations before the conduct of any study-related procedures. They must be able and willing to participate in all scheduled evaluations, abide by all study restrictions, and complete all required tests and procedures.

Exclusion criteria:

MSA group:

History of other neurological disorders or intracranial co-morbidities, such as stroke, haemorrhage, space-occupying lesions.

Presence of supranuclear gaze palsy. Presence of any clinically significant medical condition (including cardiovascular, respiratory, cerebrovascular, hematological, hepatic, renal, gastrointestinal, or other disease) that, based on the judgement of the investigator, is clinically unstable, is likely to deteriorate during the course of the study, could put the patient at risk because of participation in the study, could affect the subject's ability to complete the study, or could influence the study results.

Severe-to-complete dependence on caregivers (score >3 on UMSARS Part IV, Global Disability), severe impairment of swallowing (score ≥3 on UMSARS Part I, Question 2), or frequent falls (score ≥3 on UMSARS Part I, Question 8) at Screening.

Presence of any of the following MRI contraindications: pacemaker; cardiac defibrillator; spinal cord or vagus nerve stimulator; aneurysm clip; artificial heart valve; recent coronary or carotid stent; ear implant; CSF shunt; other implanted medical device (e.g. Swan-Ganz catheter, insulin pump); or metal fragments or foreign objects in the eyes, skin, or body. If the principal investigator considers the presence of any of the above not to be a contraindication to MRI in a given subject, the investigator may obtain approval from the MR operators based on a discussion of the case.Negative modified Allen test in both hands.

History of claustrophobia or back pain that makes prolonged laying on the MRI or PET scanner intolerable.

Pregnancy, lactation, or, if female of childbearing potential, positive urine β-hCG at screening or prior to PET scan.

Use of drugs acting on SV2A such as antiepileptics (e.g. levetiracetam or brivaracetam).

History of brain surgery for parkinsonism or stem cell treatment. Clinically significant blood clotting or bleeding disorder, including clinically significant abnormal findings in laboratory assessments of coagulation or hematology.

Current or recent history of alcohol or drug abuse / dependence (except nicotine dependence).

History of cancer within the last 5 years, with the exception of nonmetastatic basal cell carcinoma of the skin.

Hemoglobin A1c (HbA1c) ≥ 6.5% at screening. Uncontrolled/poorly controlled diabetes mellitus.

For subjects participating in optional CSF sampling:

* Any spinal malformation or other aspects (e.g. tattoos) / clinical findings (e.g. papilledema) that may complicate or contraindicate lumbar puncture, as judged by the investigator.
* Neoplasm or other space-occupying intracranial lesion on MRI. Any clinically important abnormality, as determined by the investigator, on physical examination or vital signs, ECG, or clinical laboratory test results other than abnormality due to a stable, well-controlled medical condition; or any abnormality that could be detrimental to the subject or could compromise the study.

PSP group:

History of other neurological disorders or intracranial co-morbidities, such as stroke, haemorrhage, space-occupying lesions.

Inclusion in any clinical trial with investigational drugs targeting tau. Presence of any clinically significant medical condition (including cardiovascular, respiratory, cerebrovascular, hematological, hepatic, renal, gastrointestinal, or other disease) that, based on the judgement of the investigator, is clinically unstable, is likely to deteriorate during the course of the study, could put the patient at risk because of participation in the study, could affect the subject's ability to complete the study, or could influence the study results.

Presence of any of the following MRI contraindications: pacemaker; cardiac defibrillator; spinal cord or vagus nerve stimulator; aneurysm clip; artificial heart valve; recent coronary or carotid stent; ear implant; CSF shunt; other implanted medical device (e.g. Swan-Ganz catheter, insulin pump); or metal fragments or foreign objects in the eyes, skin, or body. If the principal investigator considers the presence of any of the above not to be a contraindication to MRI in a given subject, the investigator may obtain approval from the MR operators based on a discussion of the case.

Abnormal modified Allen test in both hands. History of claustrophobia or back pain that makes prolonged laying on the MRI or PET scanner intolerable.

Pregnancy, lactation, or, if female of childbearing potential, positive urine β-hCG at screening or prior to PET scan.

History of brain surgery for parkinsonism or stem cell treatment. Clinically significant blood clotting or bleeding disorder, including clinically significant abnormal findings in laboratory assessments of coagulation or hematology.

Current or recent history of alcohol or drug abuse / dependence (except nicotine dependence).

History of cancer within the last 5 years, with the exception of nonmetastatic basal cell carcinoma of the skin.

For subjects participating in optional CSF sampling:

• Any spinal malformation or other aspects (e.g. tattoos) / clinical findings (e.g. papilledema) that may complicate or contraindicate lumbar puncture, as judged by the investigator.

Neoplasm or other space-occupying intracranial lesion on MRI. Any clinically important abnormality, as determined by the investigator, on physical examination or vital signs, ECG, or clinical laboratory test results other than abnormality due to a stable, well-controlled medical condition; or any abnormality that could be detrimental to the subject or could compromise the study.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of MSA; patients with a diagnosis of PSP
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
To measure the magnitude of longitudinal within-group change in [11C]UCB-J volume of distribution in MSA | Baseline to 12 Months
  [11C]UCB-J is a marker of synaptic damage in MSA

SECONDARY OUTCOMES:
Progression of brain glucose metabolism in MSA | Baseline to 12 Months
  Brain glucose metabolism is assessed with serial [18F]FDG PET scans at baseline and after 12-month follow-up.
To investigate differences in MRI structural, microstructural, molecular, and functional parameters in MSA patients. | Baseline to 12 Months
  Magnetic Resonance Imaging change in Magnetization Prepared Rapid Acquisition Gradient Echo [MPRAGE]
To investigate differences in structural MRI parameters in MSA patients. | Baseline to 12 Months
  Magnetic Resonance Imaging change in Magnetization Prepared Rapid Acquisition Gradient Echo [MPRAGE]
To investigate differences in iron-sensitive MRI in MSA patients. | Baseline to 12 Months
  Magnetic Resonance Imaging change in Susceptibility Weighted Imaging [SWI]
To investigate differences in quantitative iron in MSA patients. | Baseline to 12 Months
  Magnetic Resonance Imaging change in Quantitative Susceptibility Mapping [QSM]
To investigate differences in microstructural MRI parameters in MSA patients. | Baseline to 12 Months
  Magnetic Resonance Imaging change in Diffusion Tensor Imaging [DTI]
To investigate differences in neuromelanin-MRI in MSA patients. | Baseline to 12 Months
  Magnetic Resonance Imaging change in Neuromelanin-MRI
To investigate differences in perfusion MRI parameters in MSA patients. | Baseline to 12 Months
  Magnetic Resonance Imaging change in Arterial Spin Labelling [ASL]
To investigate differences in functional MRI parameters in MSA patients. | Baseline to 12 Months
  Magnetic Resonance Imaging change in resting state functional MRI [rs-fMRI]
To investigate differences in markers of neurite density on MRI in MSA patients. | Baseline to 12 Months
  Magnetic Resonance Imaging change in Neurite Orientation Dispersion and Density Imaging [NODDI]
To investigate correlations between imaging and grading of MSA in MSA patients. | Baseline to 12 Months
  Correlations between imaging measures and the grading scale UMSARS
To investigate correlations between imaging and staging of MSA in MSA patients. | Baseline to 12 Months
  Correlations between imaging measures and the staging scale Hoehn and Yahr
To investigate correlations between synaptic density, regional brain glucose metabolism, and clinical measures in MSA patients. | Baseline to 12 Months
  Correlations between imaging measures and the screening cognitive measure MoCA
To investigate correlations between imaging measures and functional scales in MSA patients. | Baseline to 12 Months
  Correlations between imaging measures and the ability scale Schwab & England
To investigate correlations between imaging measures and quality of life in MSA patients. | Baseline to 12 Months
  Correlations between imaging measures and the quality of life scale MSA QoL
To investigate correlations between imaging measures and symptoms of autonomic dysfunction in MSA patients. | Baseline to 12 Months
  Correlations between imaging measures and the autonomic symptoms scale COMPASS-31
To investigate correlations between imaging measures and symptoms of postural instability and tendency to fall in MSA patients. | Baseline to 12 Months
  Correlations between imaging measures and the balance scale ABC-16
To investigate correlations between imaging measures and symptoms of depression in MSA patients. | Baseline to 12 Months
  Correlations between imaging measures and the depression scale BDI-II
To investigate correlations between imaging measures and symptoms suggestive of depression in MSA patients. | Baseline to 12 Months
  Correlations between imaging measures and the depression scale HDRS
To investigate correlations between imaging measures and REM sleep behaviour disorder in MSA patients. | Baseline to 12 Months
  Correlations between imaging measures and the sleep scale RBD-SQ
To investigate correlations between imaging measures and presence of behavioural symptoms in MSA patients. | Baseline to 12 Months
  Correlations between imaging measures and the behavioural scale NPI
To investigate correlations between imaging measures and cognitive decline in MSA patients. | Baseline to 12 Months
  Correlations between imaging measures and the cognitive battery CANTAB
To investigate correlations between imaging measures and fluid biomarkers of inflammation in MSA patients. | Baseline to 12 Months
  Correlations between imaging measures and blood biomarkers related to neuroinflammation
To investigate correlations between imaging measures and CSF biomarkers in MSA patients. | Baseline to 12 Months
  Correlations between imaging measures and CSF biomarkers related to neuroinflammation and misfolded proteins deposition
Change in [18F]APN107 brain uptake in patients with PSP | Baseline to 12 months
  Quantification of the changes over time of [18F]APN107 brain uptake, reflective of tau deposition, in patients with PSP
Correlation between longitudinal changes in [18F]APN107 and structural changes on MRI | Baseline to 12 months
  Magnetic Resonance Imaging change in Magnetization Prepared Rapid Acquisition Gradient Echo [MPRAGE]
To investigate differences in tau pathology across MSA and PSP patients | Baseline to 12 months
  differences in the brain uptake of [18F]APN107 between MSA and PSP patients

CONTACTS AND LOCATIONS:
Overall Officials: Marios Politis, MD MSc PhD, Study Chair — University of Exeter
Locations (1):
- University of Exeter, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: No